CLINICAL TRIAL: NCT04696484
Title: Feasibility of a Goal-based Agenda Setting Intervention for Informing Conversations in Adult Cystic Fibrosis Care
Brief Title: Feasibility of a Goal-based Agenda Setting Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Glyn Jones-Elwyn, Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00047666
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Cystic Fibrosis; Chronic Disease
MeSH Terms: conditions — Cystic Fibrosis; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): coopeRATE Prompt
  Interventions: Behavioral: coopeRATE Prompt

INTERVENTIONS:
Behavioral: coopeRATE Prompt — The coopeRATE Prompt intervention is a set of two questions delivered to patients before the clinical encounter that elicit their concerns and goals. The intervention is delivered to patients online, outside the clinic setting.

SUMMARY:
This study aims to assess the feasibility of a new, brief intervention, the 'coopeRATE Prompt', for informing conversations between patients and physicians in routine tele-health and in-person adult Cystic Fibrosis (CF) care. The coopeRATE Prompt is two questions designed to elicit patients' concerns and goals to facilitate collaborative goal setting within the health care visit. This is a prospective single arm study that will be conducted at four CF care centers in the United States.

DETAILED DESCRIPTION:
Participating patients will be asked to complete two online surveys. The first survey, which includes the coopeRATE Prompt intervention questions, is completed 1-4 days before their upcoming healthcare visit. After completing this survey and before their visit, patients' intervention responses are shared with their physician and, if requested, other members of their care team. The second patient survey is completed within 24 hours after their healthcare visit. Participating clinicians are asked to complete a single online survey within one month after completion of patient data collection.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of CF
* are 18 years of age or older
* can read and write English
* have a scheduled in-person or tele-health routine CF care visit
* have access to internet and email

Exclusion Criteria:

* does not have a diagnosis of CF
* is less than 18 years of age
* cannot read and write English
* does not have a scheduled in-person or tele-health routine CF care visit
* does have access to internet and email

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Use of intervention responses with physician (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported discussion of intervention responses (concerns and goals) in the visit with physician, assessed using two items with multiple choice (single answer) format. The first item assesses how many of the patient concerns were discussed and the second item assesses how many of the patient goals were discussed. Item response options are 'None of them', 'Some of them', or 'All of them'.

SECONDARY OUTCOMES:
Intervention completion (patient-reported) | 1-4 days before the healthcare visit
  Presence of a response to each of the coopeRATE Prompt intervention questions. The coopeRATE Prompt includes two items with open-text response format.
Intervention acceptability (patient-reported) | 1-4 days before the healthcare visit
  Patient-reported intervention acceptability, assessed using an adapted version of the 4-item Acceptability of Intervention Measure (Weiner et al., 2017). Each item is rated on a 5-point scale ranging from 1 ('Completely disagree') to 5 ('Completely agree'). A respondent's total score is the mean of all item responses.
Utility of intervention (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported utility (helpfulness) of intervention, assessed using a single adapted item (Dalcin et al., 2015). The item is rated on a 5-point scale ranging from 0 ('Not at all helpful') to 4 ('Extremely helpful').
Way(s) in which intervention was helpful (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported way(s) in which intervention was helpful, assessed using a single item with multiple choice (multiple answer) format.
Initiator of discussion (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported initiator of discussion of intervention responses in the visit with physician, assessed using a single item with multiple choice (single answer) format.
Satisfaction with time spent (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported satisfaction with amount of time spent discussing intervention responses in the visit with physician, assessed using a single item with multiple choice (single answer) format.
Preference for sharing intervention responses with other team members (patient-reported) | 1-4 days before the healthcare visit
  Patient-reported preference for sharing intervention responses with other members of the care team, assessed using a single item with multiple choice (multiple response) format.
Use of intervention responses with other team members (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported discussion of intervention responses in the visit with other members of the care team, assessed using two items. The first item assesses whether intervention responses were discussed, with a multiple choice (single answer) format. The second item assesses the specific team members with whom discussions were had, with a multiple choice (multiple answer) format.
Satisfaction with intervention timing (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported satisfaction with timing of intervention delivery, assessed using a single item with multiple choice (single answer) format.
Preferred intervention timing (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported preferred timing of intervention delivery, assessed using a single item with open-text response format.
Future receipt of intervention (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported preference for receiving the intervention again in the future, assessed using a single item with multiple choice (single answer) format.
Collaborative goal setting (patient-reported) | Within 24 hours after completion of the healthcare visit
  A new 3-item patient-reported measure under evaluation to assess collaborative goal setting between a patient and physician during the health care visit. Each item is rated on a 4-point scale ranging from 0 ('Strongly disagree') to 3 ('Strongly agree'), with an additional 'Not sure' option. Scoring method is to be determined.
Shared decision-making (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported shared decision-making with physician during the health care visit, assessed using the 3-item collaboRATE measure (Elwyn et al., 2013; Barr et al., 2014). Each item is rated on a 10-point scale ranging from 0 ('No effort was made') to 9 ('Every effort was made'). Respondent's are assigned a score of 1 if every item is rated 'Every effort was made' and a score of 0 for all other response combinations.
Frequency of intervention receipt (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported frequency of receiving patient intervention responses, assessed using a single item with open-text response format.
Use of intervention responses with patients (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported frequency of use of intervention responses with patients in the visit, assessed using a single item with multiple choice (single answer) format.
Utility of intervention (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported utility (helpfulness) of intervention, assessed using a single adapted item (Dalcin et al., 2015). The item is rated on a 5-point scale ranging from 0 ('Not at all helpful') to 4 ('Extremely helpful').
Way(s) in which intervention was helpful (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported way(s) in which intervention was helpful, assessed using a single item with multiple choice (multiple answer) format.
Impact on time spent with patients (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported impact on amount of time spent with patients, assessed using a single item with multiple choice (single answer) format.
Reason(s) for not using intervention (never used) (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported reason(s) for never discussing intervention responses with patients, assessed using a single item with multiple choice (multiple answer) format.
Reason(s) for not using intervention (sometimes used) (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported reason(s) for only sometimes discussing intervention responses with patients, assessed using a single item with multiple choice (multiple answer) format.
Intervention acceptability (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported intervention acceptability, assessed using an adapted version of the 4-item Acceptability of Intervention Measure (Weiner et al., 2017). Each item is rated on a 5-point scale ranging from 1 ('Completely disagree') to 5 ('Completely agree'). A respondent's total score is the mean of all item responses.
Future use of intervention (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported preference for using the intervention with patients in the future, assessed using a single item with multiple choice (single answer) format.

OTHER OUTCOMES:
Concerns and goals (patient-reported) | 1-4 days before the healthcare visit and within 24 hours after completion of the healthcare visit
  Patient-reported concerns and goals, assessed using the coopeRATE Prompt intervention. The coopeRATE Prompt includes two items with open-text response format. Item responses are assessed in terms of concern and goal frequency and type (categorizations to be determined).
Additional intervention feedback (patient-reported) | 1-4 days before the healthcare visit and within 24 hours after completion of the healthcare visit
  Patient-reported additional intervention feedback, assessed using two items with open-text response format. Additional feedback is first assessed immediately after completing the intervention questions and again after the index healthcare visit.
Type of routine healthcare visit (patient-reported) | Within 1 month following completion of patient data collection
  Patient-reported type of routine CF care visit (e.g., in-person only, phone-only), assessed using a single item with multiple choice (single answer) format.
People seen during the visit (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported people seen (e.g., doctor, nurse) during the healthcare visit, assessed using a single item with multiple choice (multiple answer) format.
History with people seen during the visit (patient-reported) | Within 24 hours after completion of the healthcare visit
  Patient-reported history with people seen during the healthcare visit, assessed using a single item with multiple choice (single answer) format.
Additional intervention feedback (clinician-reported) | Within 1 month following completion of patient data collection
  Clinician-reported additional intervention feedback, assessed using a single item with open-text response format.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Elwyn, Principal Investigator — Dartmouth College
Locations (4):
- United States (4):
  - National Jewish Health, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
A de-identified copy of participant-level data and essential analytic code will be made available to others for research purposes, via data sharing.
Supporting Information: Analytic Code
Time Frame: The data and supporting information will be available after December 2021 and for an indefinite period of time.
Access Criteria: Requests must include sufficient justification for the data which does not duplicate any current or planned data use. All requests will be subject to Investigator approval.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Dalcin AT, Jerome GJ, Fitzpatrick SL, Louis TA, Wang NY, Bennett WL, Durkin N, Clark JM, Daumit GL, Appel LJ, Coughlin JW. Perceived helpfulness of the individual components of a behavioural weight loss program: results from the Hopkins POWER Trial. Obes Sci Pract. 2015 Oct;1(1):23-32. doi: 10.1002/osp4.6. Epub 2015 Sep 9. PMID 27668085
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354